CLINICAL TRIAL: NCT03769064
Title: Phase 1, Single-dose, Double-blind, Rand., Placebo- and Active-controlled, 4-period, 4-sequence Crossover, Proof-of-Concept Study to Evaluate Effect of Naltrexone on Abuse Potential of Methylphenidate in Healthy Recreational Stimulant Users
Brief Title: Study for Naltrexone on the Abuse Potential of Methylphenidate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Avekshan LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: AVK-001
Record Dates: First submitted 2018-10-11; First posted 2018-12-07 (Actual); Last update posted 2018-12-07 (Actual); Status verified 2018-12

CONDITIONS: Naltrexone; Methylphenidate Abuse
Keywords: ADHD; attention deficit hyperactivity disorder; stimulant
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Intervention Model Description: The study will consist of a 2-period crossover Qualification Phase (Part 1) to ensure subject eligibility for the treatment phase of the study, and a 4-period crossover Treatment Phase (Part 2) to determine the effect of concomitant administration of MPH and NTX on subjective pharmacodynamic (PD) measures of abuse, relative to MPH and placebo.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind, randomized
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Qualification Phase (Part A) (Experimental): Placebo/Methylphenidate (60 mg) on days 1 and 3
  Interventions: Drug: Placebo; Drug: Methylphenidate 60 mg
- Qualification Phase (Part B) (Experimental): Methylphenidate (60 mg)/Placebo on days 1 and 3
  Interventions: Drug: Placebo; Drug: Methylphenidate 60 mg
- Treatment Phase Sequence 4213 (Experimental): Methylphenidate 60 mg/Naltrexone 100 mg Methylphenidate 60 mg/Placebo Placebo/Placebo Methylphenidate 60 mg/Naltrexone 50 mg
  Interventions: Drug: Treatment Phase Sequence 4213
- Treatment Phase Sequence 2134 (Experimental): Methylphenidate 60 mg/Placebo Placebo/Placebo Methylphenidate 60 mg/Naltrexone 50 mg Methylphenidate 60 mg/Naltrexone 100 mg
  Interventions: Drug: Treatment Phase Sequence 2134
- Treatment Phase Sequence 1342 (Experimental): Placebo/Placebo Methylphenidate 60 mg/Naltrexone 50 mg Methylphenidate 60 mg/Naltrexone 100 mg Methylphenidate 60 mg/Placebo
  Interventions: Drug: Treatment Phase Sequence 1342
- Treatment Phase Sequence 3421 (Experimental): Methylphenidate 60 mg/Naltrexone 50 mg Methylphenidate 60 mg/Naltrexone 100 mg Methylphenidate 60 mg/Placebo Placebo/Placebo
  Interventions: Drug: Treatment Phase Sequence 3421

INTERVENTIONS:
Drug: Placebo — Potential subjects will be screened to determine their eligibility for the study within 28 days of the first dose in the Qualification Phase (i.e., Days -28 to -2). Eligible subjects will be admitted to the clinical site on Day -1 of the Qualification Phase (Part 1) and randomized on Day 1 to receive placebo and MPH (60 mg) in 1 of 2 sequences with a 48-hour washout between dose administrations (i.e., dose administration on Days 1 and 3).
  Other Names: Qualification Phase (Part A)
  Arms: Qualification Phase (Part A); Qualification Phase (Part B)
Drug: Methylphenidate 60 mg — Potential subjects will be screened to determine their eligibility for the study within 28 days of the first dose in the Qualification Phase (i.e., Days -28 to -2). Eligible subjects will be admitted to the clinical site on Day -1 of the Qualification Phase (Part 1) and randomized on Day 1 to receive placebo and MPH (60 mg) in 1 of 2 sequences with a 48-hour washout between dose administrations (i.e., dose administration on Days 1 and 3).
  Other Names: Qualification Phase (Part A)
  Arms: Qualification Phase (Part A); Qualification Phase (Part B)
Drug: Treatment Phase Sequence 4213 — Subjects will be administered single doses on Days 1, 4, 7, and 10 of the Treatment Phase.
  Other Names: Treatment 1
  Arms: Treatment Phase Sequence 4213
Drug: Treatment Phase Sequence 2134 — Subjects will be administered single doses on Days 1, 4, 7, and 10 of the Treatment Phase.
  Other Names: Treatment 2
  Arms: Treatment Phase Sequence 2134
Drug: Treatment Phase Sequence 1342 — Subjects will be administered single doses on Days 1, 4, 7, and 10 of the Treatment Phase.
  Other Names: Treatment 3
  Arms: Treatment Phase Sequence 1342
Drug: Treatment Phase Sequence 3421 — Subjects will be administered single doses on Days 1, 4, 7, and 10 of the Treatment Phase.
  Other Names: Treatment 4
  Arms: Treatment Phase Sequence 3421

SUMMARY:
The current abuse liability study aims to assess the potential for co-administration of naltrexone (NTX) to reduce the abuse potential of methylphenidate (MPH).

DETAILED DESCRIPTION:
The abuse of MPH, as a Schedule II substance, is a well-documented problem. Studies in animal models, including primates, show that high-dose MPH can produce reinforcement or reward. A number of studies suggest that the rapid elevation of MPH levels in the blood and brain that occurs following intranasal or oral administration of supra-therapeutic doses is a key requirement for development of MPH-associated euphoria, reinforcement, and addiction. The concerns about MPH abuse potential and addiction often play a role in the decision of patients, parents, or physicians who opt against treatment with MPH, despite its effectiveness. This provides an imperative for development of MPH formulations that are therapeutically potent but with lower abuse potential. Methylphenidate acts mainly through the dopaminergic system. At sufficiently high doses, MPH can also activate the mu opioid receptors (MOPR) in the brain. Recent data indicate that blockade of MOPRs by naltrexone (NTX) blocks the rewarding effects of MPH in mice. Clinical studies on the modulatory effect of NTX on dopamine release following chronic amphetamine use also support the involvement of opioid-dopamine interactions in the reinforcing and rewarding effects of amphetamine. These data support the hypothesis that NTX will block the reinforcing effect of MPH in humans.

ELIGIBILITY:
Inclusion Criteria:

1. Recreational stimulant users, defined as ≥10 lifetime non-therapeutic experiences (i.e., for psychoactive effects) with CNS stimulants (e.g., amphetamines, cocaine, MPH) and ≥1 non-therapeutic use of a CNS stimulant within the 12 weeks prior to Screening.
2. A body mass index of ≥18 to ≤34 kg/m2 at Screening.
3. In good health, as determined by medical history, PE, vital signs assessments, 12-lead ECG, and clinical laboratory evaluations.
4. A female study subject must meet one of the following criteria:

   1. If of childbearing potential - is abstinent from heterosexual intercourse or uses 2 of the accepted contraceptive regimens from at least 30 days prior to the first administration of the study medication, during the study, and for at least 30 days after the last dose of the study medication. An acceptable method of contraception includes the following:

      * Progestogen-containing hormonal contraceptives (birth control pills, injectable/implantable/insertable hormonal birth control products, transdermal patch) and use of condom with spermicide
      * Intrauterine device (without hormones)
      * Condom
      * Spermicide
   2. If of non-childbearing potential - should be surgically sterile (i.e. has undergone complete hysterectomy, bilateral oophorectomy, or tubal ligation) or in a menopausal state (at least 1 year without menses), as confirmed by follicle-stimulating hormone (FSH) levels (postmenopausal must be confirmed by the subject having a serum FSH greater than 40 mIU/mL at Screening). Females of non-childbearing potential must present a proof of postmenopausal status and/or partial or total hysterectomy; if such proof is not available, the female will be considered to be of childbearing potential.
5. A male study subject must agree to use one of the accepted contraceptive regimens during the study and for at least 90 days after the last dose of the study medication:

   1. Abstinence from heterosexual intercourse
   2. Female partner use of hormonal contraceptives (birth control pills, injectable/implantable/insertable hormonal birth control products, transdermal patch)
   3. Female partner with intrauterine device (with or without hormones)
   4. Female partner with condom with spermicide used by male study subject
   5. Female partner of non-childbearing potential
   6. Male sterilization with absence of sperm in the post-vasectomy ejaculate A male study subject must agree not to donate sperm during the study and for at least 90 days after the last dose of the study medication.
6. Subjects must agree to refrain from use of any prescription or over-the-counter medications (with the exception of stable oral, implanted, or injected contraceptive hormones) or herbal remedies and consumption of any alcohol within the exclusionary periods and throughout the study.
7. Subjects must be able to speak, read, and understand English in order to complete the study assessments.
8. Able to provide written informed consent to participate in the study, and to abide by the study restrictions.
9. Willing and able to comply with all study procedures, including a total of 15 overnight stays at the study site.

Exclusion Criteria:

1. Evidence of moderate or severe substance use disorder (excluding nicotine and/or caffeine) within the past 2 years, as defined by the DSM-V, or has a lifetime history of participation in a drug rehabilitation program (excluding past participation in tobacco smoking cessation program or previous court-mandated treatment).
2. History of opioid dependence.
3. Subject has a positive urine drug or alcohol screen upon admission into the clinic at the start of the Qualification or Treatment Phase (Day -1 of Parts 1 and 2), except for cannabinoids (delta-9-tetrahydrocannabinol [THC]), which may be seen because of the long half-life of THC and slow release from adipose tissue. If THC is positive, inclusion will be at the discretion of the Investigator. Tests with positive results may be repeated and/or subjects may be rescheduled at the Investigator's discretion.
4. Abnormal pulse rate, blood pressure, oral body temperature, or respiration rate at Screening and prior to administration of any study drug that, in the opinion of the Investigator, increases the risk to the subject of participation in the study. For these parameters, out-of-range values that are not clinically significant (as determined by the Investigator) may be repeated twice and the subject may be enrolled if at least 1 repeated value is within acceptable range.
5. Abnormal 12-lead ECG at Screening and prior to first dose of any study drug that, in the opinion of the Investigator, increases the risk to the subject of participation in the study.
6. Any clinically significant medical history that, in the opinion of the Investigator, increases the risk to the subject of participation in the study.
7. A history of a major surgical procedure within 30 days prior to the start of study drug administration (Day 1 of Part 1), or any planned surgery during the study.
8. A history of any clinically significant illness within 30 days of the start of study drug administration (Day 1 of Part 1), as determined by the Investigator.
9. History of liver disease.
10. History of narrow-angle glaucoma, based on medical history and/or subject self-reporting.
11. Presence of galactose intolerance, lactase deficiency, or glucose-galactose malabsorption.
12. Presence or history of any narrowing or blockage of the digestive system.
13. Donation of blood, platelets, or plasma within 3 months prior to Screening.
14. Presence or a history of any clinically significant neurological, gastrointestinal, renal, hepatic, cardiovascular, psychiatric, respiratory, metabolic, endocrine, hematological, or other major disorders (including a history of angioedema), as determined by the Investigator.
15. A family history of sudden death or sudden cardiac arrest, as determined by the Investigator.
16. Presence or history of any medically diagnosed, clinically significant Axis I psychiatric disorder (including bipolar disorder, mood disorder, anxiety disorder, thought disorder, any psychotic disorder).
17. Presence of acute suicidality (within 6 months of Screening), as evidenced by a positive response to Question 4 or 5 on the Columbia-Suicide Severity Rating Scale (C-SSRS), indicating active suicidal ideation with any intent to act, at Screening or Check-in for each part.
18. Lifetime history of suicidal behavior such that a determination of "yes" is made on the Suicidal Behavior section of the C-SSRS for "Actual Attempt," "Interrupted Attempt," "Aborted Attempt," or "Preparatory Acts or Behavior".
19. Subject history or family history of motor tics or a diagnosis of Tourette's syndrome.
20. History of seizures and/or epilepsy.
21. Receipt of any investigational medicinal product (IMP) or new chemical entity within 30 days or 5 half-lives (if known) of the first study drug administration (Day 1 of Part 1), whichever is longer.
22. Receipt of any medications known to chronically alter drug absorption or elimination processes (e.g., rifampin, glucocorticoids, St. John's wort) within 30 days of the first study drug administration (Day 1 of Part 1).
23. Previous use of any antidepressants, seizure medications, vasodepressors, or theophylline within 3 months prior to Screening. Use of other prescription medications (with the exception of stable oral, implanted, or injected contraceptive hormones) within 30 days before first dosing (Day 1 of Part 1), unless it is determined by the Investigator that there will be no impact on the study procedures or on subject safety.
24. Use of any over-the-counter systemic or topical medication, or vitamin or mineral supplements, within 14 days of first study drug administration (Day 1 of Part 1) unless, in the opinion of the Investigator, the medication will not interfere with study procedures or compromise safety.
25. Consumption of foods or beverages containing poppy seeds, grapefruit, or Seville oranges within 7 days of first study drug administration (Day 1 of Part 1).
26. History of, or a known allergic reaction to, any study drug excipients, or a history of multiple food/drug allergies, or any clinically significant allergic condition (excluding nonactive hay fever).
27. Any clinically significant abnormal PE finding.
28. In the opinion of the Investigator, any clinically significant abnormal laboratory safety findings at Screening and prior to first study drug administration (one repeat assessment at Screening and Check-in for Part 1 is acceptable).
29. Consumption of caffeine within 24 hours prior to Check-in for either study part.
30. Consumption of alcohol or alcohol-containing products within 24 hours prior to Check-in for either study part.
31. Participation in strenuous physical activity within 72 hours prior to Check-in for either study part (e.g., marathon runners, weight lifters).
32. Known presence of serum hepatitis, or positive serologic test for hepatitis B surface antigen, hepatitis C virus antibody, or human immunodeficiency virus (HIV) antibody.
33. Subjects who, in the opinion of the Investigator, should not participate in the study.
34. Use of any opioids within 14 days prior to the first study drug administration in the Treatment Phase.
35. Physical dependence on opioids based on a naloxone challenge test.
36. Elevated aspartate aminotransferase or alanine aminotransferase ≥1.5 x upper limit of normal.
37. History of additional risk factors for torsades de pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome).
38. QTcF >450 msec or any clinically significant abnormality on the 12-lead ECG at Screening or Check-in for each part.
39. Presence or history of hypertension of cardiovascular disease.
40. History of depressive disorder within the last 2 years prior to Screening, or Patient Health Questionnaire (PHQ)-9 score >9 at Screening or Check-in for each part, or history of other severe psychiatric disorders (e.g., anxiety, schizophrenia, or bipolar disorder), as declared by subject or as judged by the Investigator.
41. Females who are pregnant or lactating.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 94 (Actual)
Dates: Start 2018-03-27 (Actual); Primary Completion 2018-06-20 (Actual); Study Completion 2018-06-20 (Actual)

PRIMARY OUTCOMES:
Maximum Effect of Naltrexone | 70 days
  To evaluate the maximum effect of 2 doses (50 and 100 mg) of Naltrexone on the abuse potential of a single dose (60 mg) of Methylphenidate in healthy recreational stimulant users using the bipolar Visual Analogue Scale for Drug Liking.
  Visual Analogue Scale (bipolar) is an administered test where the patient assess the following.:
  • Drug Liking, Overall Drug Liking, Alertness/Drowsiness, Overall Take the Drug Again;
  The response anchors are 0 (strong disliking), 50 (neither like nor dislike), and 100 (strong liking).
  Visual Analogue Scale for Drug Liking will be determined periodically over the 8 hour period following each dose administration to assess for response to test question, "At this moment, my liking for this drug is...".

SECONDARY OUTCOMES:
Time to Maximum Effect of Naltrexone | 70 days
  Time to maximum effect.
Effect of Naltrexone | 70 days
  To evaluate the safety and tolerability of concomitant administration of Naltrexone (50 or 100 mg) and Methylphenidate (60 mg) in healthy recreational stimulant users using the unipolar Visual Analogue Scale for High.
  Visual Analogue Scale (unipolar) is an administered test where patient assesses the following:
  Good Effects, High, Bad Effects
  The response anchors are 0-100 with 0 being the least effect and 100 being the most effect.
  Visual Analogue Scale for High will be administered prior to each dose administration and periodically over the 8 hour period following each dose administration to assess for response to test question, "I am feeling high," with anchor points of 0 (no effect) and 100 (Extremely) being the most effect.
Time to Minimum Effect | 70 days
  Time to minimum effect (bipolar scales only)
Time-Average Area Under the Effect Curve | 70 days
  Time-average area under the effect curve.
Adverse Events | 70 days
  Incidence and severity of adverse events
Clinical Laboratory Abnormalities | 70 days
  Incidence of clinical laboratory abnormalities, based on hematology, clinical chemistry, and urinalysis (UA) test results.
Heart Rate Assessment via Electrocardiogram | 70 days
  Heart rate assessment will be performed using a 12-lead Electrocardiogram (ECG). Normal range is QTcF ≤ 450 msec.
  Single 12-lead ECGs will be repeated once if either of the following criteria apply:
  * QT interval corrected for heart rate using Fridericia's method (QTcF) >500 msec
  * QTcF change from the baseline (predose) is >60 msec. 12-lead ECGs evaluations may be repeated at the Investigator's (or designee's) discretion and may be performed at other times if judged to be clinically appropriate or if the ongoing review of the data suggests a more detailed assessment of ECGs is required. The Investigator (or designee) will perform a clinical assessment of each 12-lead ECG.
Heart Rate Assessment via Cardiac Telemetry | 70 days
  Patient's heart rate and rhythm will be assessed via continuous cardiac telemetry. Monitoring will be conducted on all dosing days from predose until at least 12 hours postdose.
  Normal range is QTcF ≤ 450 msec.
Supine Blood Pressure Assessment | 70 days
  Supine blood pressure (systolic/diastolic in mmHg) - normal range for measurements: systolic blood pressure - 86-140 mmHg and diastolic blood pressure - 50-90 mmHg
Supine Pulse Rate Assessment | 70 days
  Supine pulse rate (beats per minute) - normal range is 50-100 beats/minute
Respiratory Rate Assessment | 70 days
  Respiratory rate (breaths per minute) - normal range is 10-24 breaths/minute
Oral Body Temperature Assessment | 70 days
  Oral body temperature (degrees Celsius) - normal range is 36.1-37.4°C
Physical Examinations (PEs) | 70 days
  The following assessments will be performed for Physical Examinations (PEs):
  * General Appearance
  * HEENT (head, eyes, ears, nose and throat))
  * Neck/Thyroid
  * Cardiovascular
  * Respiratory
  * Gastrointestinal
  * Musculoskeletal/Extremities
  * Skin
  * Other (will be specified)
Maximum Observed Plasma Concentration | 70 days
  maximum observed plasma concentration
Time of the Maximum Observed Plasma Concentration | 70 days
  Time of the maximum observed plasma concentration
Area Under the Plasma Concentration-time Curve | 24 hours
  Area under the plasma concentration-time curve from hour 0 to 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Pradeep Bhide, PhD, Study Director — Co-Founder and Chief Scientist
Locations (1):
- Vince & Associates Clinical Research, Inc., Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: No